CLINICAL TRIAL: NCT04941716
Title: AVENUE-2: Acalabrutinib in Combination With Venetoclax (AV) for Previously Treated Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
Brief Title: Acalabrutinib in Combination With Venetoclax for the Treatment of Refractory or Recurrent Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma, The AVENUE-2 Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1121341; NCI-2021-05947 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10602 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2021-06-21; First posted 2021-06-28 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; venetoclax; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (acalabrutinib, venetoclax) (Experimental): Patients receive acalabrutinib PO BID and venetoclax PO QD on days 1-28. Patients receive acalabrutinib alone for the first three 28 day cycles. Venetoclax is added beginning with Cycle 4. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.
  Patients also undergo blood sample collection, bone marrow aspiration and biopsy, and CT or MRI throughout the trial.
  Interventions: Drug: Acalabrutinib; Drug: Venetoclax; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196; Calquence
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto
Procedure: Biospecimen Collection — Undergo blood sample collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
Procedure: Computed Tomography — Undergo CT
  Other Names: CT Scan; CAT Scan; Computed Axial Tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: MRI

SUMMARY:
This phase II trial is to evaluate the effects of acalabrutinib in combination with venetoclax in treating patients with chronic lymphocytic leukemia or small lymphocytic lymphoma that does not respond to treatment (refractory) or that has come back (recurrent). Acalabrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Chemotherapy drugs, such as venetoclax, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Given acalabrutinib and venetoclax may kill more cancer cells.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive acalabrutinib orally (PO) twice a day (BID) and venetoclax PO once daily (QD) on days 1-28. Patients receive acalabrutinib alone for the first three 28 day cycles. Venetoclax is added beginning with Cycle 4. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection, bone marrow aspiration and biopsy, and computed tomography (CT) or magnetic resonance imaging (MRI) throughout the trial.

After completion of study treatment, patients are followed-up every 12 weeks and annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Men and women >= 18 years of age.
* Diagnosis of CLL or small lymphocytic lymphoma (SLL) that meets the published diagnostic criteria.
* Active disease per IWCLL 2018 criteria that require treatment. At least one of the following:

  * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia
  * Massive (> 6 cm below left costal margin), progressive, or symptomatic splenomegaly
  * Massive nodes (> 10 cm in longest diameter), or progressive or symptomatic lymphadenopathy
  * Progressive lymphocytosis with an increase of > 50% over a 2-month period or lymphocyte-doubling time of < 6 months. Lymphocyte-doubling time may be obtained by linear regression extrapolation of absolute lymphocyte counts obtained at intervals of 2 weeks over an observation period of 2 to 3 months. In patients with initial blood lymphocyte counts of < 30 x 109/L lymphocyte-doubling time should not be used as a single parameter to define treatment indication. In addition, factors contributing to lymphocytosis or lymphadenopathy other than CLL/SLL (e.g., infection) should be excluded.
  * Constitutional symptoms, defined as any 1 or more of the following disease-related symptoms or signs

    * Unintentional weight loss of > 10% within the previous 6 months
    * Significant fatigue
    * Fevers > 100.5 degrees Fahrenheit (F) or 38 degrees Celsius (C) for 2 weeks without other evidence of infection
    * Night sweats for > 1 month without evidence of infection
* Relapsed or refractory to at least 1 prior systemic therapy for CLL/SLL. A line of therapy is defined as completing at least 2 cycles of treatment of standard regimen according to current National Comprehensive Cancer Network (NCCN) guidelines, or of an investigational regimen on a clinical trial.
* Absolute neutrophil count (ANC) >= 750 cells/microliter (0.75 x 10^9/L); ANC >= 500 cells/microliter (0.50 x 10^9/L) in subjects with documented bone marrow involvement of CLL (independent of growth factor or transfusion support within 1 week of screening).
* Hemoglobin >= 10 g/dL (independent of growth factor or transfusion support within 1 week of screening).
* Platelet count >= 50,000 cells/microliter (50 x 10^9/L); platelet count >= 25,000 cells/microliter (25 x 10^9/L) in subjects with documented bone marrow involvement of CLL (independent of growth factor or transfusion support within 1 week of screening).
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* Total bilirubin =< 2 x ULN, unless directly attributable to Gilbert's syndrome
* Estimated creatinine clearance of >= 50 mL/min
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Women of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and for 30 days after the last dose of acalabrutinib or venetoclax, whichever occurs later
* Willing and able to participate in all required evaluations and procedures in this study protocol, including swallowing capsules or tablets without difficulty
* Ability to understand the purpose and the risks of the study and provide signed and dated informed consent and authorization to use protected health information

Exclusion Criteria:

* Known prolymphocytic leukemia or history of, or currently suspected, Richter's transformation (biopsy based on clinical suspicion may be needed to rule out transformation)
* Prior disease progression while on a BTK inhibitor
* Prior disease progression while on venetoclax
* Prior intolerance to acalabrutinib or venetoclax
* Prior malignancy (or any other malignancy requiring active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, low-grade prostate carcinoma (Gleason grade =< 6) or other cancer from which the subject has been disease free for >= 2 years or which will not limit survival to < 3 years
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 or 4 cardiac diseases as defined by the New York Heart Association Functional Classification, or corrected QT interval (QTc) > 480 msec at screening. Subjects with controlled, asymptomatic atrial fibrillation during screening can enroll on study.
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass. Patients with history of such operations are eligible if in treating physician's opinion they have no absorption issues.
* Known history of drug-specific hypersensitivity or anaphylaxis to acalabrutinib or venetoclax
* Active bleeding or history of bleeding diathesis (e.g. hemophilia or von Willebrand disease), or requires/is receiving anticoagulation with warfarin or equivalent vitamin K antagonists
* Prothrombin time (PT)/international normalized ratio (INR) or activated partial thromboplastic time (aPTT) (in the absence of lupus anticoagulant) > 2 x ULN
* Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP)
* Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening
* Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor or inducers. The use of strong or moderate CYP3A inhibitors or inducers within 7 days of the first dose of study drug is prohibited.
* For patients receiving capsule formulation of acalabrutinib only: Requires treatment with proton pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole) at the time of enrollment. Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
* History of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug
* Major surgical procedure within 7 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug
* Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HBc) positive and who are surface antigen negative will need to have a negative polymerase chain reaction (PCR). Those who are hepatitis B surface antigen (HbsAg) positive or hepatitis B PCR positive will be excluded. Subjects who are hepatitis C antibody positive will need to have a negative PCR result. Those who are hepatitis C PCR positive will be excluded.
* Breastfeeding or pregnant
* Concurrent participation in another therapeutic clinical trial
* Known history of infection with human immunodeficiency virus (HIV) or any active significant infection (e.g,. bacterial, viral, or fungal)
* History of or ongoing confirmed central nervous system (CNS) CLL
* History of confirmed progressive multifocal leukoencephalopathy (PML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2027-08-10 (Estimated); Study Completion 2031-08-10 (Estimated)

PRIMARY OUTCOMES:
Rate of undetectable measurable residual disease (uMRD) | At the end of treatment (26 cycles, 1 cycle = 28 days)
  MRD will be assessed using multicolor flow cytometry (sensitivity 10^-4) (uMRD4) from peripheral blood (PB).

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 10 years
  Evaluated as defined by International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018.
Complete response (CR) | Up to 10 years
  Evaluated as defined by International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018.
Partial response (PR) | Up to 10 years
  Evaluated as defined by International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018.
Progression-free survival (PFS) | Time from receiving the first treatment to the first observation of disease progression or death from any cause, whichever occurs first, assessed up to 10 years
  Kaplan-Meier curves and median time-to-event estimation with 95% confidence intervals will be presented.
Overall survival (OS) | Time from receiving the first treatment to death from any cause, assessed up to 10 years
  Kaplan-Meier curves and median time-to-event estimation with 95% confidence intervals will be presented.
Toxicity of combination | Up to 10 years
  Defined as grade 3-4 hematologic and non-hematologic malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Mazyar Shadman, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No